CLINICAL TRIAL: NCT05840198
Title: Evaluating the Impact of a Canine-assisted Therapy Program in Youth Residing in a Residential Treatment Center.
Brief Title: LH Canine Therapy Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Canine Therapy Corps (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-1104
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-03

CONDITIONS: Emotion Regulation; Behavioral Disorder; Self Esteem
MeSH Terms: conditions — Emotional Regulation; Mental Disorders | interventions — Salvage Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): Half of youth will be assigned to the active Recovery & Care Canine-Assisted Therapy intervention arm.
  Interventions: Behavioral: Recovery & Care Canine-Assisted Therapy
- Waitlist control (Other): Half of youth will receive treatment as usual.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Recovery & Care Canine-Assisted Therapy — Active intervention. An 6-week session of structured, goal-oriented activities where youth focus on mastering dog obedience and dog training skills. Each session is 1 hour and 15 minutes in length and includes education, review of prior sessions, and specific skill-building activities. Skill-building activities progress in complexity during the course of the 6-week curriculum.
  Arms: Active intervention
Other: Treatment as usual — Youth in this condition receive treatment as usual from their health care providers
  Arms: Waitlist control

SUMMARY:
The goal of this pilot project is to test for initial efficacy of the Recovery & Care Canine-Assisted Therapy program that has been developed and implemented in youth institutionalized for behavioral and emotional problems. We are using two study sites, Lawrence Hall and Lydia Home, both Chicago-based residential treatment centers for youth with behavioral and emotional problems, many of whom have experienced child maltreatment and trauma. Comparisons will be made to a matched sample of youth from Lawrence Hall and Lydia Home receiving treatment as usual. Results from this project will provide preliminary evidence of whether a structured, goal-oriented intervention program focused on dog training activities has direct impact on increasing youth emotional self-regulation, impulse control, and self-efficacy, which are important targets for intervention among youth with mental health problems. If successful, this project could lead to a larger, randomized control clinical trials study that tests the longitudinal impact of the program that could further lead to national dissemination of the Recovery & Care curriculum as an alternative therapeutic approach.

DETAILED DESCRIPTION:
The study uses a longitudinal, within-person design with two parallel conditions. In one condition, youth receive a 6-week canine therapy intervention. The other condition consists of treatment as usual. The subject population are youth that are in a full-time residential treatment facility in Lawrence Hall and Lydia Home.

The Recovery & Care Canine-Assisted Therapy intervention is a 1.25 hour structured curriculum that will occur weekly across a period of 6 weeks. The program will be delivered by the Canine Therapy Corps (CTCorps). Youth will work with CTC-affiliate staff, including trained dog-handler teams, a canine behavior expert, and a clinical supervisor to engage in a series of structured activities progress throughout the intervention. Week 1 is a "meet-and-greet" session where youth are introduced to all dog-handler teams participating in the program and will be asked to select a team to work with for the following sessions. Each youth is assigned their own dog-handler team. Weeks 2 cover activities regarding dog obedience, building from mastering basic commands which the dog already knows (such as "sit," "stay'") to the introduction of "new tricks" that the dog has not yet learned. In Weeks 3, youth will continue to work on mastering the "new tricks" with their dog-handler team and will also begin dog agility training. The agility training session progress in terms of complexity of number and types of obstacles. Week 4 is for proofing all skills (obedience, trick, agility) learned in previous sessions. Week 5 continues proofing all skills and is discussion of the graduation structure and dress rehearsal, and Week 6 is a graduation ceremony where family and friends are invited to observe the progress each youth has made with their dog-handler team. In Weeks 1-5, the goals of each session are outlined at the beginning of the session and brief education is provided regarding the session goals. Weeks 2-5 also include a review of the skills/activities covered in prior weeks. At the end of sessions 1-5, youth are asked to reflect on what they did during the session, including discussion of what they did really well, what they wanted to work on further, and goals for the next session. Research staff will be present during all sessions to record fidelity measures. The Positive and Negative Affect Scale will be administered on-site by research staff at the beginning and end of each intervention session. Change in affect are primary and secondary outcome measures.

Baseline and Follow-up data will be collected up to 1-month before and 1-month after the intervention programs from both the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Youth must be receiving in-patient services at Lawrence Hall or Lydia Home
* Youth must provide informed assent.
* Youth must complete at least one of the primary outcomes during the baseline assessment.
* Youth must remain in residential care for the duration of the 6-week intervention.
* Youth assigned to the Recovery & Care intervention group must attend at least one of the 6 sessions.

Exclusion Criteria:

* Severe cognitive, psychiatric, or physical condition or limitation that would prevent participation.
* Severe animal allergy
* Animal phobia
* History of mistreatment of animals.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Emotional Stroop | Up to 1-month post-intervention
  Computer-Assisted task assessing affect regulation
Change in Emotional Stroop | Change from baseline to up to 1-month post-intervention
  Computer-Assisted task assessing affect regulation
Flanker Task | Up to 1-month post-intervention
  Computer-Assisted task assessing attention & inhibitory control
Change in Flanker Task | Change from baseline to up to 1-month post-intervention
  Computer-Assisted task assessing attention & inhibitory control
Rosenberg Self-Esteem Scale | Up to 1-month post-intervention
  10-item self-report scale assessing self-esteem. Higher scores are better outcomes
Change in Rosenberg Self-Esteem Scale | Change from baseline to up to 1-month post-intervention
  10-item self-report scale assessing self-esteem. Higher scores are better outcomes
Change in Negative Affect | Change from the beginning to the end of each of the 6 intervention session
  In addition to overall change in outcomes post intervention, we are also interested in whether each intervention session produces an immediate change in youth emotion. We will assess negative affect using 5 self-report items on current mood from positive and negative affect scale. Higher scores are worse outcomes.

SECONDARY OUTCOMES:
Attendance and Attrition | Aggregated across the 6-week intervention program
  Project staff will record the number of absences and drop-outs for youth enrolled in both study intervention conditions.
Change in Positive Affect | Change from the beginning to the end of each of the 6 intervention session.
  In addition to overall change in outcomes post intervention, we are also interested in whether each intervention session produces an immediate change in youth emotion. We will assess positive affect using 5 self-report items on current mood from positive and negative affect scale. Higher scores are better outcomes.
Significant Event Report | Aggregated across the 6-week intervention program
  Mandated reporting of disruptive behaviors (including offenses, aggression, running away, etc.) and disciplinary actions that occur during the course of the youth's placement at Lawrence Hall.
Change in Attitudes towards Pets | Change from baseline to up to 1-month post-intervention
  Pet-Attitudes Survey-Modified (PAS-M) is a validated, reliable 18-item instrument used to assess youth attitudes towards pets. The PAS-M will be used to determine whether the Recovery & Care intervention improves attitudes towards pets and/or whether the intervention is effective for all youth. Higher scores indicate a more positive attitude.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lawrence Hall Child & Family Treatment Center, Chicago, Illinois
  - Lydia Home, Evanston, Illinois